CLINICAL TRIAL: NCT01748383
Title: Autologous Mononuclear and Cluster of Differentiation 133+ (CD 133+) Bone Marrow Cells, Growth Factors and Cytokines in the Remodeling of the Heart in Patients During and in the Late Periods After STEMI.
Brief Title: The Long-term and Short-term Efficacy and Safety of Transplantation Autologous Bone Marrow Cells (BMCs) in Patients With the First STEMI (ST Segment Elevation Myocardial Infarction)
Acronym: ESTABOMA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Russian Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Vyacheslav Ryabov, Leading researcher of Emergency Cardiology Department, Russian Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 99
Record Dates: First submitted 2012-12-07; First posted 2012-12-12 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Vascular Diseases; Cardiovascular Diseases; Acute Myocardial Infarction
Keywords: Bone marrow cells; Acute myocardial infarction; Transplantation of autologous mononuclear; Transplantation of autologous CD133 + cells
MeSH Terms: conditions — Vascular Diseases; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Transplantation of BMMCs (Experimental): Autologous BMCs aspiration and transplantation of these cells
  Interventions: Procedure: Transplantation of BMMCs
- Transplantation of CD 133+ cells (Experimental): Autologous CD 133+ BMCs aspiration and transplantation of CD 133+ cells
  Interventions: Procedure: Transplantation of CD 133+ cells
- stenting of IRA (Active Comparator): The only stenting of IRA
  Interventions: Procedure: stenting of IRA

INTERVENTIONS:
Procedure: Transplantation of BMMCs — The wing of the ilium was punctured under the local anesthesia for receiving of autologous BMCs. 100 ml of bone marrow aspirate was taken. BMMCs were obtained by the method of the gradient centrifugation. Autologous BMMCs in the number 93±43 million transplantation by balloon catheter performed into IRA at once after stent implantation.
  Arms: Transplantation of BMMCs
Procedure: Transplantation of CD 133+ cells — The wing of the ilium was punctured under the local anesthesia for receiving of autologous BMCs. 100 ml of bone marrow aspirate was taken. Autologous CD133 + cells were obtained by the method of the magnetic separation. Phenotyping of the transplanted cells was performed by the cytofluorimetry. Autologous CD 133+ BMCs in the number 5,7 (0,45;9,0) million transplantation by balloon catheter performed into IRA at once after stent implantation.
  Arms: Transplantation of CD 133+ cells
Procedure: stenting of IRA — The only stent implantation
  Arms: stenting of IRA

SUMMARY:
The purpose of this study is to test the hypothesis that the intracoronary transplantation of autologous mononuclear and CD 133 + bone marrow cells will improve left ventricular contractile function and will reduce the combined end points after the primary STEMI (mortality, recurrent myocardial infarction, angina, heart failure, stroke).

DETAILED DESCRIPTION:
The study was randomized, opened, controlled. 85 patients with the first STEMI were enrolled. Patients were divided to three groups. On admission all patients were received thrombolytic therapy by 1,5 million U streptokinase. Transplantation of autologous mononuclear bone marrow cells (BMMCs) and аutologous CD133 + cells by balloon catheter placed into infarct-related artery (IRA) was performed at once after stent implantation in 28 patients patients (1st group) and in 10 patients (2nd group) on the 7-21 days of STEMI. Another 47 patients (3nd group) undergo only stent implantation into IRA the same day of STEMI.

Autologous BMMCs were obtained from bone marrow aspirate by gradient centrifugation. Echocardiography, Holter monitoring were performed. Plasma concentration of the pro-inflammatory and anti-inflammatory cytokines (IL1, 6,8,10), of the growth factors (stem cell factor - SCF, vascular endothelial growth factor - VEGF, hepatocyte growth factor - HGF, fibroblast growth factor - FGF, insulin-like growth factor - IGF), the number of circulating CD34 +38-, CD133 +, СD117 +, CD90 +34- stem cells were determined in these patients in the acute and sub-acute myocardial infarction period.

It is going 7 years after the beginning of planned to evaluate left ventricular function of these patients, incidence of cardiovascular end points (death, recurrent myocardial infarction, angina, heart failure, stroke) and their combinations, to evaluate the safety of transplantation of autologous BMCs (formation of intra-myocardial tumor or neoplastic processes of other sites) after 7 years from the beginning of study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and to 75 Years
* Informed consent
* First STEMI
* Term admission to an intensive care unit in the first 24 hours of onset
* Time reperfusion of the IRA is not earlier than 4 hours after the initial onset of acute transmural myocardial infarction

Exclusion Criteria:

* Atrial fibrillation, a permanent form Valvular heart disease
* Severe comorbidity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2005-09; Primary Completion 2013-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Left ventricular ejection fraction (Echo) | for an average of 7 years

SECONDARY OUTCOMES:
incidence of cardiovascular death | 7 years
incidence of the recurrent myocardial infarction | 7 years
incidence of the angina | 7 years
incidence of the heart failure | 7 years
incidence of the stroke | 7 years
incidence of the combined endpoint | 7 years
incidence and severity of adverse events | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Vyacheslav Ryabov, MD, PhD, Principal Investigator — Scientific and Research Institution of Cardiology of Siberian Department of RAMS
Locations (1):
- Scientific and Research Institution of Cardiology of Siberian Department of RAMS, Tomsk, Russia